CLINICAL TRIAL: NCT05616897
Title: Physiological Responses During a 30 Minutes Sustained CPR Sequence With Feedback in Female Rescuers: a Comparison Between Medicine and Physical Education Students.
Brief Title: Physiological Responses During Sustained CPR.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B670201112158
Record Dates: First submitted 2015-02-10; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Sustained CPR

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medicine students (Other): students with normal expected fitness
  Interventions: Behavioral: Physiological responses during sustained CPR
- Physical education students (Other): students with better expected fitness
  Interventions: Behavioral: Physiological responses during sustained CPR

INTERVENTIONS:
Behavioral: Physiological responses during sustained CPR

SUMMARY:
Background Since fatigue seems related to poorer physical fitness rather than to gender, we analyzed the physiological responses during a 30 minutes sustained CPR sequence.

Methods and results Handgrip strength and VO2 max determined strength and endurance. Twenty-three medicine (M) and 27 physical education (PE) female students performed 30 minutes CPR. Compression quality and ECG were continuously monitored, heartrate and non-invasive blood pressure (NIBP) every 2 minutes. Capillary pH, PcCO2, lactate, potassium and sodium bicarbonate were analyzed every 10 minutes.

DETAILED DESCRIPTION:
2.1. Data collection Fifty female students who completed a CPR course in accordance with the 2010 ERC Guidelines were recruited on a voluntary base at the faculty of Medicine and Health Sciences (Ghent University, Belgium). Given the reports of several authors that the physical characteristics of the rescuers (including gender) had no impact on their CPR performance, we did not use a male control group. This prospective data collection was carried out at Ghent University Hospital and approved by the research Ethics Committee (B670201112158) and informed consent was obtained from every participant.

2.2 Study protocol The participants were divided into two groups according to their expected physical condition: Medicine students (M; n=23) and Physical Education students (PE; n=27). As a consequence of their curriculum we expected the physical education students to have a good or at least better physical condition compared to the medical students. The participants' height (anthropometer GPM, DKSH Switzerland), weight (electronic SECA, 815 Elegantia) and body fat percentage (Harpende Skinfold Calliper, Fysio Supplies) were measured. Body mass index (BMI; kg/m²) was calculated. To assess baseline strength and endurance respectively, we measured hand grip strength (kg) (Hydraulic hand dynamometer, Sachon corporation, Mason) as a determinant of general muscle strength and we estimated maximal oxygen uptake (ml/kg/min) by means of an endurance shuttle run test as a parameter of maximal aerobic power.In order to detect unknown cardiac abnormalities a 12 lead ECG (Delta 60 plus, Cardioline) was performed in all volunteers.

All participants were considered as lay rescuers and had received previous CPR training. However, to avoid any pre-testing difference, each group received a CPR instruction booster, using the ERC-accredited 4-stage approach, one week before the study.

After this, the students were asked to perform a 30 minutes sustained CPR sequence (30:2). Regarding the available evidence on the impact of CPR feedback devices on CPR quality, participants were given real-time feedback on hand positioning, compression depth, ventilation volume and a metronome continuously provided a rhythm of 100-120 compressions per minute.(5) CPR quality data were registered using a Laerdal Resusci Anne manikin (Laerdal, Norway) connected to a Laerdal PC Skill reporting software (version 2.4) and simultaneously monitored by an observer.

To define compressions as adequate, they were automatically evaluated for depth (>5 cm), frequency (100-120/min) and complete release (<0.5 cm). The ventilations were automatically evaluated for the inflated volume (400-1000 ml). The 30:2 CPR was performed during 30 minutes with a hands-off period every 2 minutes during the AED analysis. This time interval was used to measure and register the volunteers heart rate (bpm), non-invasive blood pressure (NIBP) and peripheral oxygen saturation (SpO2), which was repeated every 2 minutes. All participants were connected to a continuous 5 lead ECG monitor (SC 9000 xl, Siemens). In addition to the non invasive monitoring, capillary blood samples from the fingertip were taken every 10 minutes to analyze the pH, PcCO2, lactate, potassium and sodium bicarbonate (Radiometer ABL90 Flex, Denmark). The results of the non-invasive and capillary monitoring were evaluated by an anaesthesiologist and exercise physiologist throughout the whole exercise. In case of hypertension or arrhythmia, tiredness, feeling unwell or failure to maintain correct compression rhythm or depth the participant was asked to stop the physical effort and the reason was noted. At the end of the 30 minutes the participants were asked to appraise their feeling of exertion on a "Borg rating of perceived exertion scale" ranging from 6 to 20.

ELIGIBILITY:
Inclusion Criteria:

Medicine or Physical education student

Exclusion Criteria:

hypertension arrhythmia failure to maintain correct compression rhythm or depth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Difference in blood pressure between female medicine and physical education students during a 30 minutes sustained CPR sequence. | 30 minutes
Difference in heart rate between female medicine and physical education students during a 30 minutes sustained CPR sequence. | 30 minutes
Difference in respiration rate between female medicine and physical education students during a 30 minutes sustained CPR sequence | 30 minutes
Difference in pCO2 between female medicine and physical education students during a 30 minutes sustained CPR sequence. | 30 minutes
Difference in pO2 between female medicine and physical education students during a 30 minutes sustained CPR sequence. | 30 minutes
Difference in lactate values between female medicine and physical education students during a 30 minutes sustained CPR sequence. | 30 minutes